CLINICAL TRIAL: NCT07162051
Title: A Single-arm, Open-label Study of Fluzoparib Combination With Chemotherapy for Neoadjuvant Treatment of HRD-positive, HR+/HER2- Breast Cancer
Brief Title: A Study on the Use of Fluzoparib Combined With Chemotherapy for Neoadjuvant Treatment of HRD-positive, HR+/HER2- Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20222031-F-2
Record Dates: First submitted 2025-08-14; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: HR+/HER2- Early Breast Cancer
Keywords: Fuzaparib; breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Flutaparib combined with standard chemotherapy (Experimental): Subjects will receive fluzoparib combined with docetaxel followed by epirubicin and cyclophosphamide. After fully understanding the study and signing the informed consent form, eligible subjects identified by researchers will enter the trial period. The trial drug must be administered within 72 hours after confirmation of enrollment. Each treatment cycle lasts 3 weeks, with a total of 8 cycles. In cycles 1-4, subjects receive fluzoparib combined with docetaxel; in cycles 5-8, they receive epirubicin and cyclophosphamide. Administration continues until the end of the treatment course, or until disease progression, occurrence of intolerable toxicity, or withdrawal of informed consent by the subject.
  Interventions: Drug: Fuzaparib; Other: standard chemotherapy

INTERVENTIONS:
Drug: Fuzaparib — Folfoxapril:
  Take 2 times a day (once in the morning and once in the evening, 150mg in the morning and 100mg in the evening; vice versa is also acceptable). Each 3-week period constitutes one cycle. For the first to fourth cycles, a total of 4 cycles are required.
Other: standard chemotherapy — standard chemotherapy

SUMMARY:
The purpose of this clinical trial is to evaluate the efficacy and safety of Fluzoparib combined with docetaxel in sequential paclitaxel combined with cyclophosphamide for HRD-positive, HR+/HER2- early breast cancer. The main question it aims to answer is:

Does the proportion of patients with residual tumor burden (RCB) 0/I increase when Fluzoparib combined with docetaxel is sequentially followed by paclitaxel combined with cyclophosphamide for patients with HRD-positive, HR+/HER2- early breast cancer? What medical problems will participants encounter when using Fluzoparib combined with docetaxel in sequential paclitaxel combined with cyclophosphamide?

Participants will:

After confirming their enrollment, they need to receive the trial drug treatment within 72 hours, with each 3-week period as a treatment cycle, for a total of 8 cycles. The first to fourth cycles will receive Fluzoparib combined with docetaxel treatment, and the fifth to eighth cycles will receive paclitaxel and cyclophosphamide treatment. The treatment will continue until the end of the treatment course or disease progression, occurrence of intolerable toxicity, or the subject withdrawing the informed consent form.

DETAILED DESCRIPTION:
This study is a single-arm, exploratory clinical trial, which plans to enroll 28 eligible subjects with HRD-positive, ER-positive, HER2-negative early breast cancer. They will receive fluzoparib combined with standard chemotherapy, aiming to observe and evaluate the efficacy and safety of fluzoparib combined with docetaxel followed by epirubicin and cyclophosphamide in the treatment of HRD-positive, HR+/HER2- early breast cancer.

Subjects will receive fluzoparib combined with docetaxel followed by epirubicin and cyclophosphamide. After fully understanding the study and signing the informed consent form, eligible subjects identified by researchers will enter the trial period. The trial drug must be administered within 72 hours after confirmation of enrollment. Each treatment cycle lasts 3 weeks, with a total of 8 cycles. In cycles 1-4, subjects receive fluzoparib combined with docetaxel; in cycles 5-8, they receive epirubicin and cyclophosphamide. Administration continues until the end of the treatment course, or until disease progression, occurrence of intolerable toxicity, or withdrawal of informed consent by the subject.

This study is conducted in 3 phases: screening phase, treatment phase, and follow-up phase.

* Screening Phase

  * Collect basic information of subjects (including date of birth, gender, ethnicity, etc.);
  * Researchers will inquire about and record in detail the subject's medical history (including past medical history and current medical history) as well as drug allergy status. The doctor may require the subject to provide relevant records of diagnosis and treatment in other hospitals, so please cooperate to provide them;
  * Check the subject's blood pressure, pulse, body temperature, and respiratory rate;
  * Tumor diagnosis: date of pathological confirmation, pathological type, pathological stage (TNM), clinical stage.
  * Tumor treatment history

    * History of tumor surgery: name of surgery, date of surgery;
    * History of radiotherapy: radiotherapy site, dose, start and end dates;
    * History of concomitant diseases, past medication history, drug allergy history, etc.;
  * Comprehensive physical examination: general condition, head and face, skin, lymph nodes, eyes, ears, nose and throat, oral cavity, respiratory system, cardiovascular system, abdomen, reproductive-urinary system, musculoskeletal system, nervous system, and mental state, etc.
  * Vital signs: pulse, respiratory rate, body temperature, and blood pressure.
  * ECOG score.
  * Blood routine: red blood cell count (RBC), hemoglobin (Hb), platelet count (PLT), white blood cell count (WBC), neutrophil count (ANC), lymphocyte count.
  * Blood biochemistry: including Glucose, TP, ALT, AST, ALP, γ-GT, ALB, TBIL, TG, CHOL, BUN, etc.
  * Urine routine: white blood cells, red blood cells, urine protein.
  * Coagulation function
  * Virological tests: HBsAg, HBsAb, HBeAg, HBeAb, HBcAb (qualitative; if HbsAg is positive, HBV DNA quantitative detection must be performed), HCV-Ab (if positive, HCV-RNA quantitative detection must be performed), and HIV-Ab.
  * 12-lead electrocardiogram: at least heart rate, QT, QTc, and P-R intervals must be indicated.
  * Echocardiogram: at least left ventricular ejection fraction (LVEF) must be indicated. It should be performed within 28 days before the first administration.
  * Imaging examinations: imaging examinations of the head, neck, chest, abdomen, pelvis, and bone tissue (such as enhanced MRI of the head, enhanced CT scans of the chest, upper abdomen, and pelvis, whole-body bone scan, etc.).
  * Tumor tissue samples: pathological tissue samples and peripheral blood samples need to be provided before enrollment for HRD and BRCA mutation detection.
  * Clinical breast examination (CBE) (including breast/axilla/supraclavicular fossa), breast ultrasound and/or mammography, and magnetic resonance imaging (MRI) scan;
  * Before neoadjuvant therapy, physical marking of tumor lesions must be performed in accordance with the standard clinical operation specifications of the research center (such as skin tattooing or surgical metal clips, etc.).
  * If the subject's clinical and/or ultrasound examination suggests axillary lymph node metastasis, axillary staging should include fine needle aspiration (FNA) or core needle biopsy before neoadjuvant therapy.
* Treatment Phase

After participating in the trial, subjects will receive fluzoparib combined with docetaxel followed by epirubicin and cyclophosphamide as determined by researchers until disease progression. The contents and steps to be evaluated during the trial include:

ECOG score, vital signs, blood routine, urine routine; blood biochemistry; 12-lead electrocardiogram, echocardiogram, tumor imaging examinations, adverse events, recording of concomitant medications and concomitant treatments; breast surgery, surgical diagnosis and treatment of axillary lymph nodes; postoperative case evaluation; diagnosis of recurrence or reoccurrence.

During each visit, the doctor will inform you of the time and place of the next visit. Throughout the study treatment process, subjects need to fill in the "Medication Diary Card" every day to record their medication status, as well as any uncomfortable symptoms and concomitant medications during this period.

·Follow-up Phase

When subjects complete the study treatment or terminate the study treatment early due to intolerable toxicity or other reasons, they need to go to the hospital to complete an exit study follow-up. The researcher will arrange the following examination items:

Physical examination: blood routine, urine routine, blood biochemistry, and coagulation function will be completed; Electrocardiogram examination: 12-lead electrocardiogram; Recording of adverse events; Recording of concomitant medications/concomitant treatments.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following inclusion criteria to be enrolled in this trial:

1. Female patients with newly diagnosed breast cancer, aged ≥18 years and ≤70 years;
2. Histopathologically confirmed early or locally advanced HR+/HER2- invasive breast cancer, as defined by the latest ASCO/CAP guidelines, meeting the following conditions:

   * HER2-negative: IHC 0/1+ or IHC 2+ with negative ISH;
   * ER-positive: IHC >1%; PR-positive: IHC >1%;
   * cT1c or above with positive lymph nodes; cT2 or above with negative lymph nodes must meet at least one of the following: age ≤40 years; Ki67 >50%; lymphovascular invasion; histological grade III;
   * HRD-positive: defined as HRD score ≥42 points and/or germline BRCA1/2 mutation (pathogenic or likely pathogenic);
   * ECOG performance status 0-1;
3. Presence of at least one measurable lesion according to RECIST 1.1 criteria;
4. Organ function must meet the following requirements:

1) Hematology

* Absolute neutrophil count (ANC) ≥1.5×109/L (no use of hematopoietic stimulating factors within 14 days before the first administration of the study drug);
* Platelet count (PLT) ≥100×109/L (no blood transfusion within 14 days before the first administration of the study drug);
* Hemoglobin (Hb) ≥90 g/L; 2) Blood biochemistry
* Total bilirubin (TBIL) ≤1.5×ULN;
* Aspartate transaminase and alanine transaminase (ALT and AST) ≤2.5×ULN;
* Blood urea nitrogen (BUN) and creatinine (Cr) ≤1.5×ULN; 3) Cardiac function
* Echocardiogram: LVEF ≥50%;
* 12-lead electrocardiogram: QTc interval <470 ms in females. 5. Subjects voluntarily participate in the study and sign the informed consent form.

Exclusion Criteria

Subjects with any of the following conditions are excluded:

1. Tumor-related symptoms and treatment 1) Patients with metastatic breast cancer or bilateral breast cancer; 2) Patients with inflammatory breast cancer; 3) Participation in other drug trials or receipt of any anti-tumor therapy (including endocrine therapy, bisphosphonate therapy, immunotherapy, biological therapy, or tumor embolization) within 4 weeks before enrollment; 4) Previous treatment with PARP inhibitors;
2. Comorbidities/medical history 1) Previous history of other malignant tumors that have received any systemic anti-tumor therapy or local treatment (including surgery and radiotherapy), excluding cured malignant tumors such as carcinoma in situ of the cervix, basal cell carcinoma, or squamous cell carcinoma; 2) Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome; active hepatitis (hepatitis B, defined as HBV-DNA ≥500 IU/ml; hepatitis C, positive anti-HCV and HCV-RNA above the lower limit of detection by the analytical method) or combined hepatitis B and C co-infection; autoimmune hepatitis; 3) Severe infection within 4 weeks before the first administration, including but not limited to bacteremia requiring hospitalization, severe pneumonia, etc.; or active infection of CTCAE ≥Grade 2 requiring systemic antibiotic treatment within 2 weeks before the first administration, or unexplained fever >38.5°C during screening/first administration (fever caused by tumors, as judged by the investigator, is allowed); 4) Subjects with a history of or planned allogeneic bone marrow transplantation or solid organ transplantation; 5) Severe heart disease or disorders, including but not limited to:

   * Confirmed history of heart failure or systolic dysfunction (LVEF <50%);
   * High-risk uncontrolled arrhythmias, such as atrial tachycardia with resting heart rate >100 bpm, significant ventricular arrhythmias (e.g., ventricular tachycardia), or high-grade atrioventricular block (i.e., Mobitz II second-degree or third-degree atrioventricular block);
   * Angina pectoris requiring anti-anginal medication;
   * Clinically significant valvular heart disease;
   * ECG showing transmural myocardial infarction;
   * Poorly controlled hypertension (systolic blood pressure >180 mmHg and/or diastolic blood pressure >100 mmHg);
3. Pregnant or lactating women, women of childbearing potential with positive baseline pregnancy test, or women of childbearing potential unwilling to use effective contraception throughout the trial period;
4. Previous clear history of neurological or psychiatric disorders, including epilepsy or dementia; known history of psychiatric drug abuse, alcoholism, or drug addiction;
5. Any other conditions deemed inappropriate for the study by the investigator.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-03-03 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Residual tumor burden (RCTB) 0/I | Two weeks after the surgery

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | up to 24 weeks
Event-free survival time (EFS) | maybe 10 years after the surgery
  EFS is calculated from the start of chemotherapy until the first detection of tumor recurrence, disease progression, or death-whichever comes first.
Overall Survival (OS) | Ten years after the surgery or even longer
  OS is defined as the duration from the starting point to death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided